CLINICAL TRIAL: NCT04148560
Title: Validity of the Remote Food Photography Method to Measure Food Intake in Adolescents in Free-living Conditions
Brief Title: Free-living Validation of the RFPM in Adolescents
Acronym: FoodPhone2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 2019-053
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Dietary Assessment; Energy Intake; Food Intake; Food Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study sample (Other): Individuals who participate in this validation study
  Interventions: Other: Tests of the validity of the RFPM and SmartIntake app.

INTERVENTIONS:
Other: Tests of the validity of the RFPM and SmartIntake app. — Participants who enroll will be trained in using the RFPM/SmartIntake app and a food record and will complete the Food Intake Assessment Preference Survey. They will also use both methods to estimate intake during a simulated lab-based meal (they will not eat during this simulated meal). They will be dosed with DLW at this visit and will use the RFPM for the subsequent 1-2 days to get accustomed to using the method, with the following three days comprising the data collection period.

SUMMARY:
The primary aim of this small study is to test the validity of the Remote Food Photography Method and an updated SmartIntake app in a sample of adolescents. The investigators will test the validity (accuracy) of the method/app at estimating energy intake in free-living conditions over approximately three days compared to doubly labeled water. This is a small study that has low statistical power, but will provide important data nonetheless and inform future research.

DETAILED DESCRIPTION:
Energy intake (EI) is an important predictor of weight gain (1) and accurate methods to measure children's and adolescent's EI are needed. Self-report methods (e.g., 24-hour recall and food records) have their strengths and are frequently used to measure children's EI. Nonetheless, they also have significant limitations, including participant and caregiver burden and lack of near real-time data.

Our group developed the Remote Food Photography Method (RFPM) to measure the EI of adults in near real-time and the validity data in adults are exceptional; the RFPM underestimates EI in laboratory settings by less than 6% and in free-living conditions by less than 7% compared to weighed foods and by less than 4% compared to doubly labeled water (DLW) over 6 days. At the same time, participant burden is drastically reduced compared to self-report methods, as participants are only required to capture images of their food selection and plate waste with a smartphone app and send these images to the laboratory for analysis. This validation study aims to assess the accuracy of the RFPM and SmartIntake app in a sample of adolescents in free-living conditions.

ELIGIBILITY:
Inclusion Criteria:

* boy or girl of any race
* age between 12 and 18 years
* willingness to use the RFPM/SmartIntake app for 3 days, in addition to a 1-2 day run-in period
* willingness to be responsive to study staff when prompted for additional information when using the RFPM/SmartIntake app
* parental support of the project, except for 18-year-olds

Exclusion Criteria:

* Individuals may not qualify for this study based on other eligibility criteria not listed. The study coordinator determine this on a case-by-case basis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Equivalence between energy intake (kcal/day) measured with the RFPM and DLW | 3 days
  Energy intake is measured by the RFPM and DLW in kcal per day over 3 days. We will use the mean of the 3 days in the analyses. Two one-sided paired t-tests (α = 0.05 for each) will be performed in this pilot with equivalence bounds at 2% increments between 8% and 34% to determine equivalence in kcal estimates between RFPM and DLW.

SECONDARY OUTCOMES:
Mean difference between the RFPM and DLW on kcal/day | 3 days
  RFPM - DLW (kcal), with each method measuring energy intake over three days, and the mean of the three days for each method being included in the calculations and analyses.
Mean percentage error of RFPM relative to DLW | 3 days
  MPE = (RFPM - DLW) / DLW × 100

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Access to individual de-identified data is possible via Pennington Biomedical Research Center's Data Sharing policy.